CLINICAL TRIAL: NCT02626052
Title: Diagnostic Accuracy of the Vibration Induced Nystagmus Test in Room Light.
Brief Title: Helpfulness of the Vibration Test Performed in Room Light on Clients With Inner Ear Problems
Status: Completed | Type: Observational
Sponsor: Aultman Health Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 2015.11.19.F1
Record Dates: First submitted 2015-12-01; First posted 2015-12-10 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Vestibular Disease
Keywords: Skull vibration induced nystagmus test; mastoid vibration test
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Dizziness Handicap Inventory — A standardized questionnaire used to quantify symptoms of dizziness.
Behavioral: Global Rating of Change — A standardized questionnaire used to review the overall outcome of the participants condition with physical therapy.
Behavioral: Patient Acceptable Symptom State — A standardized questionnaire used to determine whether meaningful progress has been made
Procedure: Spontaneous Nystagmus Test — An observational test procedure used to identify involuntary eye movements caused by inner ear and/or brain dysfunction. The test is performed both in room light and with fixation blocked with a Micromedical Technologies infrared lens.
Procedure: Gazehold Nystagmus Test — An observational test procedure used to identify involuntary eye movements caused by inner ear and/or brain dysfunction. The test is performed both in room light and with fixation blocked with a Micromedical Technologies infrared lens.
Procedure: Primary Vibration Test — A test used to identify asymmetry that may be present in the vestibular system through 60-100 MHz vibration applied to the mastoid bone. A WAHL massager is used to stimulate the inner ear by vibrating the mastoid bone. The test is performed both in room light and with fixation blocked with a Micromedical Technologies infrared lens.

SUMMARY:
The purpose of this study is to explore the diagnostic values associated with both a positive and negative Skull Vibration Induced Nystagmus Test (SVINT) performed in room light (with fixation). The hypotheses include: 1. A positive room light SVINT will be identified in individuals with moderate to severe vestibular asymmetries. 2. A positive room light SVINT will be present when 10 beats or more (counted over 10 seconds) of nystagmus are found with fixation blocked.

DETAILED DESCRIPTION:
Dizziness and vertigo account for about four million visits to the Emergency Department per year and costs for management in the Emergency Department are estimated to be about four billion dollars per year. Vestibular problems are a major cause of dizziness. Simple to perform and inexpensive bedside vestibular tests are needed. The Skull Vibration-Induced Nystagmus Test (SVINT) with fixation blocked has been considered a vestibular gold standard test with strong psychometric values. No studies on the diagnostic accuracy of the SVINT in room light have been performed.

ELIGIBILITY:
Inclusion Criteria:

* Clients 18 years and older with complaint of dizziness, vertigo, and/or imbalance who are willing to proceed with procedures of study.
* Inclusion for control group: no history of dizziness, vertigo, and/or imbalance.

Exclusion Criteria:

* Conditions that warrant immediate referral to the Emergency Department or Primary Care Physician (undiagnosed and unstable disorders relating to cardiac, neurologic, metabolic, etc, dysfunction); no history of dizziness, vertigo, and/or balance problems.
* Clients with conditions that therapists believe may be aggravated by testing including, but not limited to: variants of head injuries, migraines, seizure disorders, panic/anxiety, claustrophobia, severe headache and/or nausea, and hypersensitivity to sensory stimuli

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with complaints of dizziness, vertigo, and/or imbalance referred to the hospital outpatient physical therapy department.
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2015-12; Primary Completion 2017-01-26 (Actual); Study Completion 2017-01-26 (Actual)

PRIMARY OUTCOMES:
Primary Vibration Test | Baseline
  Under room light, the presence or absence of nystagmus is determined. If nystagmus is present, then the direction of nystagmus is determined. When fixation is blocked, the presence or absence of nystagmus is determined. If nystagmus is present, then the direction of nystagmus is determined. The number of beats per 10 sec is also determined.

SECONDARY OUTCOMES:
Dizziness Handicap Inventory | Baseline; last day of physical therapy, an average of 4 weeks
  Score on DHI.
Global Rating of Change | Baseline; last day of physical therapy, an average of 4 weeks
  Score on Global Rating of Change
Patient Acceptable Symptom State | Baseline; last day of physical therapy, an average of 4 weeks
  Yes or No response
Spontaneous Nystagmus Test | Baseline
  Presence, intensity, and direction of nystagmus is determined
Gazehold Nystagmus Test | Baseline
  Presence, intensity, and direction of nystagmus is determined

CONTACTS AND LOCATIONS:
Overall Officials: Andy Beltz, PT, Principal Investigator — Aultman Health Foundation